CLINICAL TRIAL: NCT01844518
Title: A Phase 3 Multi-center, Open-Label Study to Evaluate Pharmacokinetics, Efficacy and Safety of Abatacept Administered Subcutaneously (SC) in Children and Adolescents With Active Polyarticular Juvenile Idiopathic Arthritis (pJIA) and Inadequate Response (IR) to Biologic or Non Biologic Disease Modifying Anti-rheumatic Drugs (DMARDs)
Brief Title: Pharmacokinetics, Efficacy and Safety of Abatacept Administered Subcutaneously (SC) in Children and Adolescents With Active Polyarticular Juvenile Idiopathic Arthritis (pJIA) and Inadequate Response (IR) to Biologic or Non Biologic Disease Modifying Anti-rheumatic Drugs (DMARDs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-301; 2012-003195-39 (EudraCT Number)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Active Polyarticular Juvenile Idiopathic Arthritis
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Short and Long Terms: Orencia (Experimental): Short Term: Orencia 50 mg/mL, 87.5 mg/mL, 125 mg/mL pre-filled syringes subcutaneously (0.4 mL/0.7 mL/1.0 mL) weekly for 4 months
  Long term: Orencia 50 mg/mL, 87.5 mg/mL, 125 mg/mL pre-filled syringes subcutaneously (0.4 mL/0.7 mL/1.0 mL) weekly for 20 months
  Interventions: Biological: Abatacept

INTERVENTIONS:
Biological: Abatacept
  Other Names: Orencia

SUMMARY:
The purpose of this study is to estimate Abatacept steady-state trough concentration (Cmin) at Day 113 in children and adolescents with pJIA

ELIGIBILITY:
Inclusion Criteria:

* JIA subjects (male or female), ages 2-17 years with active disease who had an insufficient therapeutic response or intolerance to at least one non biologic DMARD or Tumor Necrosis Factor (TNFα) antagonists for at least 3 months prior to screening
* Subjects with TNFα inadequate response (or prior biologic) will be restricted to 30% of the population
* Subjects must have a history of at least 5 joints with active disease and must have currently active articular disease with ≥2 active joints and ≥2 joints with limitation of motion.

Exclusion Criteria:

* Subjects with other rheumatic diseases or major chronic inflammatory/immunologic diseases, active uveitis, systemic JIA with active systemic features (within a period of 6 months prior to enrollment), persistent Oligoarthritis JIA, or failed 3 or more TNFα antagonists or other biological DMARDs will be excluded.
* Active systemic disease: (ie, extra-articular features of systemic JIA including fever, rash, organomegaly) within a period of 6 months prior to randomization.
* Subjects who have failed more than two TNFα antagonists or other biologic DMARDs

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2015-03-12 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (57):
- United States (12):
  - Local Institution - 0007, Birmingham, Alabama
  - Local Institution - 0003, Little Rock, Arkansas
  - Local Institution - 0011, Hartford, Connecticut
  - Local Institution - 0009, Chicago, Illinois
  - Riley Hospital For Children, Indianapolis, Indiana
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Local Institution - 0001, Kansas City, Missouri
  - Local Institution - 0002, The Bronx, New York
  - Local Institution - 0008, Cincinnati, Ohio
  - Local Institution - 0005, Portland, Oregon
  - Local Institution - 0004, Salt Lake City, Utah
  - Seattle Children'S Hospital, Seattle, Washington
- Argentina (5):
  - Local Institution - 0029, Rosario, Santa Fe Province
  - Local Institution - 0028, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0030, Buenos Aires
  - Local Institution - 0064, CABA
  - Local Institution - 0031, Córdoba
- Belgium (3):
  - Local Institution - 0037, Brussels
  - Local Institution - 0036, Ghent
  - Local Institution - 0049, Leuven
- Brazil (5):
  - Local Institution, Curitiba, Paraná
  - Local Institution - 0038, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0042, São Paulo
  - Local Institution - 0040, São Paulo
  - Local Institution - 0041, São Paulo
- France (5):
  - Local Institution - 0018, Bron
  - Local Institution - 0016, Le Kremlin-Bicêtre
  - Local Institution - 0014, Paris
  - Local Institution - 0017, Poitiers
  - Local Institution - 0015, Strasbourg
- Germany (5):
  - Local Institution - 0044, Bad Bramstedt
  - Local Institution - 0045, Berlin
  - Local Institution - 0046, Hamburg
  - Local Institution - 0048, Heidelberg
  - Local Institution - 0047, Sankt Augustin
- Italy (4):
  - Local Institution - 0061, Florence
  - Local Institution, Genova
  - Local Institution - 0022, Milan
  - Local Institution - 0062, Napoli
- Mexico (5):
  - Local Institution - 0060, Guadalajara, Jalisco
  - Local Institution - 0059, Mexico City, Mexico City
  - Local Institution - 0057, Mexico City, Mexico City
  - Local Institution - 0056, Monterrey, Nuevo León
  - Local Institution - 0058, Mérida, Yucatán
- Peru (4):
  - Local Institution - 0027, Lima
  - Local Institution, Lima
  - Local Institution - 0025, Lima
  - Local Institution - 0026, Lima
- Local Institution - 0068, Tolyatti, Russia
- South Africa (4):
  - Local Institution - 0035, Park West, Bloemfontein, Free State
  - Local Institution - 0032, Pretoria, Gauteng
  - Local Institution - 0034, Pretoria, Gauteng
  - Local Institution - 0033, Cape Town, Western Cape
- Spain (4):
  - Local Institution - 0050, Barcelona
  - Local Institution - 0053, Madrid
  - Local Institution - 0055, Madrid
  - Local Institution - 0052, Valencia

REFERENCES:
- [Derived] Ruperto N, Lovell DJ, Berman A, Anton J, Viola DO, Lauwerys B, Rama ME, Bohnsack J, Breedt J, Fischbach M, Lutz T, Minden K, Ally M, Rubio-Perez N, Gervais E, Van Zyl R, Wong R, Askelson M, Martini A, Brunner HI; Pediatric Rheumatology Collaborative Study Group (PRCSG) and the Paediatric Rheumatology International Trials Organisation (PRINTO). Abatacept as Monotherapy and in Combination With Methotrexate in Patients With Juvenile Idiopathic Arthritis: Analysis of 2 Phase III Trials. J Rheumatol. 2023 Nov;50(11):1471-1480. doi: 10.3899/jrheum.2022-1320. Epub 2023 Jul 15. PMID 37453737
- [Derived] Brunner HI, Tzaribachev N, Louw I, Calvo Penades I, Avila-Zapata F, Horneff G, Foeldvari I, Kingsbury DJ, Paz Gastanaga ME, Wouters C, Breedt J, Wong R, Askelson M, Zhuo J, Martini A, Lovell DJ, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG) investigators. Long-Term Maintenance of Clinical Responses by Individual Patients With Polyarticular-Course Juvenile Idiopathic Arthritis Treated With Abatacept. Arthritis Care Res (Hoboken). 2023 Nov;75(11):2259-2266. doi: 10.1002/acr.25156. Epub 2023 Jun 22. PMID 37221146
- [Derived] Ruperto N, Lovell DJ, Berman A, Avila-Zapata F, Horneff G, Alessio M, Becker ML, Belot A, Burgos-Vargas R, Gamir ML, Goldenstein-Schainberg C, Scheibel IM, Terreri MT, Zemel L, Zhuo J, Askelson M, Wong R, Martini A, Brunner HI; Pediatric Rheumatology Collaborative Study Group and the Paediatric Rheumatology International Trials Organisation. Patient-Reported Outcomes Among Patients Ages Two to Seventeen Years With Polyarticular-Course Juvenile Idiopathic Arthritis Treated With Subcutaneous Abatacept: Two-Year Results From an International Phase III Study. Arthritis Care Res (Hoboken). 2023 Aug;75(8):1804-1814. doi: 10.1002/acr.24989. Epub 2023 Jan 29. PMID 36710243
- [Derived] Ruperto N, Brunner HI, Tzaribachev N, Vega-Cornejo G, Louw I, Cimaz R, Dare J, Espada G, Faugier E, Ferrandiz M, Gerloni V, Quartier P, Silva CA, Wagner-Weiner L, Gandhi Y, Passarell J, Nys M, Wong R, Martini A, Lovell DJ; Pediatric Rheumatology Collaborative Study Group (PRCSG) and the Paediatric Rheumatology International Trials Organisation (PRINTO). Absence of Association Between Abatacept Exposure and Initial Infection in Patients With Juvenile Idiopathic Arthritis. J Rheumatol. 2021 Jul;48(7):1073-1081. doi: 10.3899/jrheum.200154. Epub 2021 Jan 15. PMID 33452173
- [Derived] Brunner HI, Tzaribachev N, Cornejo GV, Joos R, Gervais E, Cimaz R, Calvo Penades I, Cuttica R, Lutz T, Quartier P, Gandhi Y, Nys M, Wong R, Martini A, Lovell DJ, Ruperto N; Pediatric Rheumatology Collaborative Study Group and the Paediatric Rheumatology International Trials Organisation. Maintenance of antibody response to diphtheria/tetanus vaccine in patients aged 2-5 years with polyarticular-course juvenile idiopathic arthritis receiving subcutaneous abatacept. Pediatr Rheumatol Online J. 2020 Feb 22;18(1):19. doi: 10.1186/s12969-020-0410-x. PMID 32087715
- [Derived] Brunner HI, Tzaribachev N, Vega-Cornejo G, Louw I, Berman A, Calvo Penades I, Anton J, Avila-Zapata F, Cuttica R, Horneff G, Foeldvari I, Keltsev V, Kingsbury DJ, Viola DO, Joos R, Lauwerys B, Paz Gastanaga ME, Rama ME, Wouters C, Bohnsack J, Breedt J, Fischbach M, Lutz T, Minden K, Miraval T, Ally MMTM, Rubio-Perez N, Solau Gervais E, van Zyl R, Li X, Nys M, Wong R, Banerjee S, Lovell DJ, Martini A, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Subcutaneous Abatacept in Patients With Polyarticular-Course Juvenile Idiopathic Arthritis: Results From a Phase III Open-Label Study. Arthritis Rheumatol. 2018 Jul;70(7):1144-1154. doi: 10.1002/art.40466. Epub 2018 May 20. PMID 29481737
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 219 participants were treated.
Groups:
- SC Abatacept Ages 6 to 17: Subcutaneous (SC) abatacept administered by prefilled syringe (PFS) once weekly according to the following weight-tiered dosing regimen: 10 to less than (<) 25 kilogram (kg) (50 milligram [mg] in 0.4 milliliter [mL] PFS), 25 to < 50 kg (87.5 mg in 0.7 mL PFS) and 50 kg (125 mg in 1 mL PFS).
- SC Abatacept Ages 2 to 5: SC abatacept administered by PFS once weekly according to the following weight-tiered dosing regimen: 10 to < 25 kg (50 mg in 0.4 mL PFS), 25 to < 50 kg (87.5 mg in 0.7 mL PFS) and 50 kg (125 mg in 1 mL PFS).
Period: Overall Study
Arm/Group | SC Abatacept Ages 6 to 17 | SC Abatacept Ages 2 to 5
Started | 173 | 46
Completed | 132 | 39
Not Completed | 41 | 7
Not completed — Adverse Event | 7 | 1
Not completed — Lack of Efficacy | 17 | 5
Not completed — Participant's request to discontinue | 4 | 1
Not completed — Poor/Non-compliance | 1 | 0
Not completed — No Longer Met Study Criteria | 2 | 0
Not completed — Withdrawal by Subject | 9 | 0
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated population included all participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | SC Abatacept Ages 6 to 17 | SC Abatacept Ages 2 to 5 | Total
Number analyzed (Participants) | 173 | 46 | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 173 | 46 | 219
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 28 | 164
  Male | 37 | 18 | 55
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    Black or African American | 14 | 1 | 15
    White | 144 | 44 | 188
    More than one race | 0 | 0 | 0
    Other | 15 | 1 | 16
Weight [Count of Participants; unit: Participants]
  <25 kg | 18 | 43 | 61
  25 to 50 kg | 74 | 3 | 77
  >=50 kg | 81 | 0 | 81

OUTCOME MEASURES:

1. Primary Outcome: Abatacept Trough Concentration (Cmin) in Participants Ages 6 to 17
Description: Trough concentration of abatacept (reported as geometric mean of Cmin) in all pharmacokinetic (PK)-evaluable participants. Cmin is reported in microgram per milliliter (µg/mL). Desired target therapeutic Cmin should be >= 10 µg/mL.
Time Frame: Day 113
Population: All treated participants with available PK measurements. Endpoint pre-specified to only be collected for 6-17 year age group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | SC Abatacept Ages 6 to 17
Number analyzed (Participants) | 131
µg/mL | 39.7 (35)

2. Secondary Outcome: Percentage of Participants (Ages 6 to 17) Achieving American College of Rheumatology Pediatric 30 Response (ACRp30)
Description: ACRp30 is defined as ≥30% improvement in at least 3 of the 6 juvenile idiopathic arthritis (JIA) core set variables:
  1. number of active joints
  2. number of joints with limitation of motion (LOM)
  3. physician global assessment of disease activity
  4. parent global assessment of patient overall well-being
  5. functional ability as measured by the Children's Health Assessment Questionnaire (CHAQ)
  6. C-reactive protein (CRP). In addition to the above condition, to be considered a responder participants cannot have ≥30% worsening in more than 1 of the 3 remaining JIA core set variables for which improvement was not observed.
Time Frame: Day 113
Population: All treated participants in the 6-17 Year Age-Group Cohort. Endpoint prespecified to only be collected for 6-17 year age group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SC Abatacept Ages 6 to 17
Number analyzed (Participants) | 173
Percentage of participants | 83.2 [77.7 to 88.8]

3. Secondary Outcome: Abatacept Trough Concentration (Cmin) in Participants Ages 6 to 17 by Weight Tier Dose
Description: Evaluation of the trough concentration of abatacept (reported as geometric mean of Cmin) in all pk-evaluable participants at Days 57, 85 and 113. Weight-tiered dosing groups are based on the first dose the participant received. Cmin is reported in microgram per milliliter (µg/mL). Here 'n' number analyzed signifies participants who were evaluable for each time point.
Time Frame: Days 57, 85 and 113
Population: All treated participants with available PK measurements in the 6-17 Year Age-Group Cohort. Endpoint pre-specified to only be collected for 6-17 year age group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Groups:
- 10 to <25 kg Dosing Group: Weight-tiered dosing group received 50 mg SC abatacept administered to 6 to 17 year old participants by PFS once weekly.
- 25 to <50 kg Dosing Group: Weight-tiered dosing group received 87.5 mg SC abatacept administered to 6 to 17 year old participants by PFS once weekly.
- >=50 kg Dosing Group: Weight-tiered dosing group received 125 mg SC abatacept administered to 6 to 17 year old participants by PFS once weekly
Arm/Group | 10 to <25 kg Dosing Group | 25 to <50 kg Dosing Group | >=50 kg Dosing Group
Number analyzed (Participants) | 17 | 69 | 74
microgram per milliliter (µg/mL)
  Day 57: number analyzed (Participants) | 14 | 69 | 74
  Day 57 | 29.5 (32) | 36.2 (35) | 33.0 (33)
  Day 85: number analyzed (Participants) | 17 | 63 | 65
  Day 85 | 27.7 (38) | 42.5 (32) | 36.0 (40)
  Day 113: number analyzed (Participants) | 15 | 61 | 55
  Day 113 | 34.3 (39) | 44.2 (34) | 36.6 (31)

4. Secondary Outcome: Number of Participants With Adverse Events (AEs), Deaths, Serious AEs (SAEs) and AEs Leading to Discontinuation in the Short-Term Period for the 6-17 Year Age-Group Cohort
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational product, whether or not considered related to the investigational product. A SAE is any untoward medical occurrence that at any dose which results in death, is life threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect.
Time Frame: From first dose up to 56 days post last dose in the short-term period (initial 4-month treatment period)
Population: All treated participants in the short-term period in the 6-17 Year Age Group Cohort. Endpoint pre-specified to only be collected for 6-17 year age group.
Measure: Count of Participants; unit: Participants
Arm/Group | SC Abatacept Ages 6 to 17
Number analyzed (Participants) | 173
Participants
  Deaths | 0
  SAEs | 5
  Drug-Related SAEs | 1
  Discontinuation due to SAEs | 2
  Overall AEs | 102
  Drug-Related AEs | 36
  Discontinuation due to AEs | 3

5. Secondary Outcome: Number of Participants With Adverse Events (AEs), Deaths, Serious AEs and AEs Leading to Discontinuation in the Cumulative Period
Description: as for outcome 4
Time Frame: From first dose up to 56 days after last dose ( up to approximately 2 years)
Population: All treated participants in the cumulative period
Measure: Count of Participants; unit: Participants
Arm/Group | SC Abatacept Ages 6 to 17 | SC Abatacept Ages 2 to 5
Number analyzed (Participants) | 173 | 46
Participants
  Deaths | 0 | 0
  SAEs | 14 | 5
  Drug-Related SAEs | 1 | 2
  Discontinuation Due to SAEs | 4 | 0
  Overall AEs | 152 | 44
  Treatment-Related AEs | 54 | 30
  Discontinuation Due to AEs | 7 | 1

6. Secondary Outcome: Number of Participants With Positive Immunogenicity Response in the Short-Term Period for the 6-17 Year Age-Group Cohort
Description: Overall number of participants with either a positive immunogenicity response for 'CTLA4 and possibly Ig' or 'Ig and/or Junction Region' relative to baseline. Sample draws for immunogenicity were scheduled at specific study days while on treatment for all subjects and at follow-up visits 28, 85, and 168 days after the last abatacept dose for those subjects who discontinued from the short term (ST) period (initial 4-month treatment period) or completed the ST study without continuing abatacept treatment.
Time Frame: From first dose up to start of LT (for those continuing in long-term) or up to 168 days after the lost dose of study medication in the ST period (for those not entering in the long-term)
Population: All treated participants in the short-term period with available immunogenicity measurements in the 6-17 Year Age-Group Cohort. Endpoint pre-specified to only be collected for 6-17 year age group.
Measure: Count of Participants; unit: Participants
Arm/Group | SC Abatacept Ages 6 to 17
Number analyzed (Participants) | 171
Participants | 3

7. Secondary Outcome: Number of Participants With Positive Immunogenicity Response in the Cumulative Period
Description: Overall number of participants with either a positive immunogenicity response for 'CTLA4 and possibly Ig' or 'Ig and/or Junction Region' relative to baseline. Sample draws for immunogenicity were scheduled at specific study days while on treatment for all subjects and at follow-up visits 28, 85, and 168 days after the last abatacept dose regardless of whether they discontinued early in the short term (ST) or long term (LT) period, elected not to enter the LT period, or completed both ST and LT periods.
Time Frame: From first dose up to 6 months following treatment discontinuation (up to approximately 2 years)
Population: All treated participants in the cumulative period with available immunogenicity measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | SC Abatacept Ages 6 to 17 | SC Abatacept Ages 2 to 5
Number analyzed (Participants) | 172 | 46
Participants | 8 | 7

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of their randomization until study completion (assessed up to approximately 113 months). SAEs and Other AEs were assessed from first dose to 168 days after last dose of study therapy (assessed up to approximately 113 months).
Description: Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | SC Abatacept Ages 6 to 17 | SC Abatacept Ages 2 to 5
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/46
Serious Adverse Events (participants affected / at risk) | 18/173 | 6/46
Other Adverse Events (participants affected / at risk) | 127/173 | 44/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SC Abatacept Ages 6 to 17 (N=173) | SC Abatacept Ages 2 to 5 (N=46)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Complicated appendicitis (Infections and infestations) | 1 | 0
Latent tuberculosis (Infections and infestations) | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Ovarian germ cell teratoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SC Abatacept Ages 6 to 17 (N=173) | SC Abatacept Ages 2 to 5 (N=46)
Anaemia (Blood and lymphatic system disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 16 | 6
Aphthous ulcer (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 2 | 3
Dental caries (Gastrointestinal disorders) | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 21 | 7
Vomiting (Gastrointestinal disorders) | 13 | 7
Pyrexia (General disorders) | 22 | 15
Bronchitis (Infections and infestations) | 12 | 4
Conjunctivitis (Infections and infestations) | 10 | 6
Gastroenteritis (Infections and infestations) | 19 | 9
Impetigo (Infections and infestations) | 3 | 4
Influenza (Infections and infestations) | 12 | 3
Molluscum contagiosum (Infections and infestations) | 3 | 3
Nasopharyngitis (Infections and infestations) | 63 | 20
Otitis media (Infections and infestations) | 3 | 3
Pharyngitis (Infections and infestations) | 11 | 6
Pneumonia (Infections and infestations) | 3 | 3
Rhinitis (Infections and infestations) | 13 | 8
Scarlet fever (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 12 | 3
Tonsillitis (Infections and infestations) | 9 | 5
Tooth abscess (Infections and infestations) | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 37 | 12
Urinary tract infection (Infections and infestations) | 11 | 2
Varicella (Infections and infestations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 3
Headache (Nervous system disorders) | 25 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.